CLINICAL TRIAL: NCT03423199
Title: Asian, International, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial of Tamoxifen With or Without Palbociclib ± Goserelin in Women With Hormone Receptor-Positive, HER2-Negative Advanced or Metastatic Breast Cancer
Brief Title: PAlbociclib Plus Tamoxifen for the Treatment of Hormone Receptor-positive, HER2-negative Advanced Breast Cancer Women - Asian studY
Acronym: PATHWAY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Pfizer (Industry); Korean Cancer Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCCH1607; WI217662 (Other: Pfizer)
Record Dates: First submitted 2018-01-09; First posted 2018-02-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms
Keywords: breast Cancer; palbociclib (PD-0332991); tamoxifen; goserelin; any menopausal status; hormone receptor positive; HER2 negative; locally advanced; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — palbociclib; Tamoxifen; Goserelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Palbociclib + Tamoxifen ± Goserelin (Experimental): Palbociclib 125 mg/day, orally once daily on Day 1 to Day 21 followed by 7 days off treatment for each 28 day cycle, plus tamoxifen 20 mg orally once daily (continuously)
  Interventions: Drug: Palbociclib; Drug: Tamoxifen; Drug: Goserelin
- Placebo + Tamoxifen ± Goserelin (Active Comparator): Placebo orally once daily on Day 1 to Day 21 followed by 7 days off treatment for each 28 day cycle, plus tamoxifen 20 mg orally once daily (continuously)
  Interventions: Drug: Placebo; Drug: Tamoxifen; Drug: Goserelin

INTERVENTIONS:
Drug: Palbociclib — Palbociclib, 125mg, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Other Names: PD-0332991
  Arms: Palbociclib + Tamoxifen ± Goserelin
Drug: Placebo — Placebo, orally once daily on Day 1 to Day 21 of every 28-day cycle followed by 7 days off treatment
  Arms: Placebo + Tamoxifen ± Goserelin
Drug: Tamoxifen — Tamoxifen, 20mg, orally once daily (continuously)
Drug: Goserelin — For pre/perimenopausal patients only: Goserelin, 3.6 mg, subcutaneously every 4 weeks; or 10.8 mg, subcutaneously every 12 weeks

SUMMARY:
This study is conducted to evaluate the benefit of adding palbociclib in hormone receptor (HR)-positive, HER2-negative advanced or metastatic breast cancer patients, regardless of menopausal status, treated with tamoxifen (with or without goserelin) versus tamoxifen alone (with or without goserelin).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older with histologically or cytologically proven locally advanced or metastatic breast cancer, not amenable to resection or radiation therapy with curative intent
* Documented diagnosis of HR+/HER2- breast cancer
* Any menopausal status
* Previously untreated with any endocrine therapy for their HR+/HER2- advanced breast cancer; or progressed while on or within 3 month from prior endocrine therapy other than tamoxifen for advanced breast cancer. If patients have adjuvant endocrine therapy, they must satisfy as follows: progressed 12 months or more since prior adjuvant endocrine therapy with tamoxifen; or progressed during or after adjuvant endocrine therapy with an aromatase inhibitor.
* Measurable disease or non-measurable disease as defined by RECIST ver.1.1
* Eastern Cooperative Oncology Group (ECOG) PS 0-1
* Adequate organ and marrow function, resolution of all toxic effects of prior therapy or surgical procedures

Exclusion Criteria:

* Prior treatment with any CDK inhibitor, tamoxifen, everolimus, or agent that inhibits the PI3K-mTOR pathway
* Patients with extensive advanced/metastatic, symptomatic visceral disease, or known uncontrolled or symptomatic CNS metastases
* Use of strong or moderate CYP3A4 and/or CYP2D6 inhibitors or inducers
* Major surgery or any anti-cancer therapy within 2 weeks of randomization
* Prior stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-02-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Baseline up to 3.5 years
  The time from the date of randomization to the date of the first documentation of objective progression of disease (PD), clinically diagnosed symptomatic deterioration, or death due to any cause in the absence of documented PD, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the randomization of the last patient up to 3 years
  The time from date of randomization to date of death due to any cause.
Survival Probabilities at 1 year, 2 year, and 3 year | From the randomization of the last patient up to 3 years
  The probability of survival 1 year, 2 or 3 years after the date of randomization based on the Kaplan-Meier estimate.
Objective Response (OR) | Baseline up to 3.5 years
  Complete response (CR) or partial response (PR) according to Response Evaluation Criteria In Solid Tumors (RECIST) ver.1.1 recorded from randomization until disease progression or death due to any cause.
Duration of Response (DR) | Baseline up to 3.5 years
  The time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death due to any cause, whichever occurs first.
Clinical Benefit Response (CBR) | Baseline up to 3.5 years
  CR or PR or SD >=24 weeks according to the RECIST version 1.1 recorded in the time period between randomization and disease progression or death of any cause.
Change From Baseline Between Treatment Comparison in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Functional Scale Scores | Baseline up to 3.5 years
  The EORTC-QLQ-C30 is a 30-item questionnaire composed of five multi-item functional subscales (physical, role, emotional, cognitive , and social functioning), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global quality of life (QOL) subscale, and six single item symptom scales assessing other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, and the financial impact of cancer). The questionnaire employs 28 4-point Likert scales with responses from "not at all" to "very much" and two 7-point Likert scales for global health and overall QOL. Responses to all items are then converted to a 0 to 100 scale. For functional and global QOL scales, higher scores represent a better level of functioning/QOL. For symptom-oriented scales, a higher score represents more severe symptoms. A 10-point or higher change in scores from baseline is considered clinically significant.
Change From Baseline Between Treatment Comparison in European Organization for Research and Treatment of Cancer Breast Cancer Module (EORTC QLQ BR23) Functional Scale Scores | Baseline up to 3.5 years
  The EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual functioning, sexual enjoyment, future perspective) and four symptom scales (systemic side effects, breast symptoms, arm symptoms, upset by hair loss). QLQ-BR23 questionnaire employs 4-point scales with responses from 'not at all' to 'very much'. All scores are converted to a 0 to 100 scale. For functional scales, higher scores represent a better level of functioning.
Trough plasma concentrations of palbociclib | Cycle 1/Day 15 and Cycle 2/Day 15
  Ctrough for palbociclib
Trough plasma concentrations of tamoxifen, 4-hydroxytamoxifen, N-desmethyltamoxifen and endoxifen | Cycle 2/Day 15 and Cycle 3/Day 15
  Ctrough for tamoxifen, 4-hydroxytamoxifen, N-desmethyltamoxifen and endoxifen
Treatment-Emergent Adverse Events | From the first dose of the investigational product until 28 days after the last dose of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Kan Yonemori, MD, PhD, Study Chair — Department of Breast and Medical Oncology, National Cancer Center Hospital
Locations (23):
- Japan (12):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Toranomon Hospital, Minato-Ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Kyusyu Cancer Center, Fukuoka
  - National Hospital Organization Osaka National Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Soeul
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Vetarans General Hospital, Taipei
  - Sun Yat-Sen Cancer Center, Taipei

REFERENCES:
- [Derived] Noguchi E, Yamanaka T, Mukai H, Yamamoto N, Chung CF, Lu YS, Chang DY, Sohn J, Kim GM, Lee KH, Lee SC, Iwasa T, Iwata H, Watanabe K, Jung KH, Tanabe Y, Kang SY, Yasojima H, Aogi K, Tokunaga E, Sim SH, Yap YS, Matsumoto K, Tseng LM, Umeyama Y, Sudo K, Kojima Y, Hata T, Kuchiba A, Shibata T, Nakamura K, Fujiwara Y, Tamura K, Yonemori K. A phase 3 study (PATHWAY) of palbociclib plus tamoxifen in patients with HR-positive/HER2-negative advanced breast cancer. NPJ Breast Cancer. 2024 Aug 22;10(1):76. doi: 10.1038/s41523-024-00684-w. PMID 39174547